CLINICAL TRIAL: NCT06744036
Title: Effects of Including Interferential Current in a Therapeutic Exercise Program in Individuals With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7.267.733
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator will only participate in the evaluation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic Exercise Group (Active Comparator): The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises.
  Interventions: Other: Therapeutic Exercise
- Therapeutic Exercises Group + Interferential Current (Experimental): The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises. However, the interferential current will be applied at the end of the therapeutic exercises. In this way, the IC will be used through a device (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square), will be positioned around the center of the knee. The parameters used were as follows: carrier current frequency of 4000 Hz; amplitude modulated frequency of 50 Hz; sweep frequency of 50 Hz; oscillation pattern of 1:1 second, and the amplitude of the current will be increased until the research participants report strong but comfortable and non-painful stimulation paresthesia. The IC will be applied for 30 minutes.
  Interventions: Other: Therapeutic Exercise; Device: Interferential Current
- Therapeutic Exercises + placebo interferential current (ET + placebo IC) group (Placebo Comparator): The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises. However, the interferential current will be applied at the end of the therapeutic exercises. In this way, the IC will be used through a device (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square), will be positioned around the center of the knee.The device will only be turned on for the first minute.
  Interventions: Other: Therapeutic Exercise; Device: placebo interferential current

INTERVENTIONS:
Other: Therapeutic Exercise — The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises.
Device: Interferential Current — However, the interferential current will be applied at the end of the therapeutic exercises. In this way, the IC will be used through a device (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square), will be positioned around the center of the knee. The parameters used were as follows: carrier current frequency of 4000 Hz; amplitude modulated frequency of 50 Hz; sweep frequency of 50 Hz; oscillation pattern of 1:1 second, and the amplitude of the current will be increased until the research participants report strong but comfortable and non-painful stimulation paresthesia. The interferential current will be applied for 30 minutes.
  Arms: Therapeutic Exercises Group + Interferential Current
Device: placebo interferential current — However, the interferential current will be applied at the end of the therapeutic exercises. In this way, the IC will be used through a device (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square), will be positioned around the center of the knee. The parameters used were as follows: carrier current frequency of 4000 Hz; amplitude modulated frequency of 50 Hz; sweep frequency of 50 Hz; oscillation pattern of 1:1 second, and the amplitude of the current will be increased until the research participants report strong but comfortable and non-painful stimulation paresthesia. The device will only be turned on in the first minute
  Arms: Therapeutic Exercises + placebo interferential current (ET + placebo IC) group

SUMMARY:
The first-line treatment for knee osteoarthritis (KOA) in terms of pain and functionality is physical exercise. The use of interferential current (IC) associated with other resources may be beneficial in reducing pain intensity and improving functionality. However, the effects of its simultaneous use with therapeutic exercise have not yet been fully established. The aim of this project will be to evaluate the effects of including IC in a therapeutic exercise program in relation to pain intensity, functionality, self-efficacy, maximum voluntary contraction and overall perceived effect in individuals with KOA. Therefore, research participants of both sexes, between 40 and 75 years old, with a clinical diagnosis of unilateral KOA, who have knee pain for more than 3 months, with a minimum score of 3 points on the numerical pain scale, morning stiffness for less than 30 minutes, crepitation, bone sensitivity and absence of palpable heat will be recruited. The research participants will be randomized into three groups: therapeutic exercises (n=42) and therapeutic exercises + IC (n=42) and therapeutic exercises + IC placebo. Eight consecutive weeks of treatment will be carried out. The research participants will be evaluated before the intervention, after the end of the intervention of eight consecutive weeks of intervention and after four weeks at the end of the last week of intervention, through the instruments: numeric pain scale (NPS), Knee Injury and Osteoarthritis Outcome Score (KOOS), patient-specific functional scale (EFEP), Pain self-efficacy questionnaire (PSEQ), maximum voluntary isometric contraction (MVIC), 30-second sit-to-stand test (TSL30s), global perception scale (EPG). For data analysis, a normality test will be used to verify the distribution of the data and a statistical test appropriate for the appropriate intra and inter-group comparisons, thus considering two factors in the comparisons, time and group. A significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* between 40 years old and 75 years old
* with a clinical diagnosis of unilateral KOA
* Who has had knee pain for more than 3 months
* With a minimum score of 3 points on the numerical pain scale
* Morning stiffness for less than 30 minutes
* Crepitus
* Bone tenderness and absence of palpable heat

Exclusion Criteria:

* Hip OA
* Severe osteoporosis
* Fibromyalgia
* Clinical history of tumors or cancer
* Active inflammatory joint diseases (rheumatoid arthritis, gout)
* Undergoing any joint replacement in the lower extremity
* Neurological diseases (Parkinson's disease, stroke
* Multiple sclerosis
* muscular dystrophies
* Diseases involving motor neurons
* Alzheimer's disease
* Infected wounds or osteomyelitis in the knee region
* Deep vein thrombosis or thrombophlebitis
* Sensory alteration in the lower limbs
* Cognitive and cardiopulmonary impairment that may prevent or limit the execution of exercises
* Use of a walking assistance device
* History of recent knee trauma
* Having undergone any form of treatment involving physical therapy
* intra-articular corticosteroids
* anti-inflammatory drugs
* opioid medication or chondroprotective in the six months before the start of the interventions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.

SECONDARY OUTCOMES:
Functional disability | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  Knee Injury and Osteoarthritis Outcome Score (KOOS). It aims to evaluate the domains of pain, symptoms, activities of daily living, function related to recreation and sports, and quality of life related to the knee. Totaling 42 items, each item must be answered using a Likert scale that ranges from 0 (best score) to 4 (worst score), and the score for each subscale ranges from 0 (worst score) to 100 (best score).
Functional self-perception | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  Pain self-efficacy questionnaire, structured into 10 items where each item is evaluated by selecting a number on a 7-point numerical scale (scores from 0 to 6), where 0 means "not at all confident" and 6 means "completely confident". The items cover different functions, from work, social activities, domestic tasks and coping with pain without medication. A total score is calculated from the sum of the scores for each of the 10 items, producing a total score that ranges from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Functional capacity | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  Sit and stand test. The volunteer will sit down and stand up from a chair for 30 seconds. A researcher will time the total time it takes to complete this activity.
Inability | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  Patient-specific functional scale. The participant will indicate three activities that he/she has difficulty performing. For each of these activities, the participant will indicate a score from 0 to 10. Higher scores indicate how well the participant can perform the activity. Lower scores indicate an inability to perform the activity.
Maximum voluntary isometric contraction | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  manual dynamometer portable (Lafayette Manual Muscle System, Modelo 01165, Lafayette Instrument Company, Lafayette, IN). Four 5-second readings will be taken during maximal voluntary isometric contraction (MVIC) with a 30-second rest period between contractions. The first CIVM will familiarize the volunteer with carrying out the task. A new set of readings will be taken if a volunteer can perform three contractions with at least 10% variability. Strong and constant verbal stimuli will be used throughout the test. Always with the research participants' hands positioned crossed on the chest. Thus, bilateral assessments of the muscles, quadriceps, and gluteus medius will be carried out. The order of CIVM readings will be randomized to avoid collection bias. The research participant will remain in lateral decubitus with a pillow positioned between the legs, with the limb to be tested superiorly in a neutral position.
Global Perception of Change scale | before the first treatment session, after 8 weeks of treatment and 4 weeks after the end of the last session
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change scale. The Global Perception of Change scale is a direct scale on the patient's self-perception when the intervention is performed. This scale consists of 11 points, ranging from -5 (worsening compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No